CLINICAL TRIAL: NCT06471270
Title: Validation of Salivary Proteomic Biomarkers for Early Detection of Oral Cancer in Egyptian Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: British University In Egypt (Other)
Responsible Party: Principal Investigator, Dalia Ghalwash, PROFESSOR, British University In Egypt
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: BU1612
Record Dates: First submitted 2024-06-14; First posted 2024-06-24 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Oral Cancer
MeSH Terms: conditions — Mouth Neoplasms | interventions — Physical Examination

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- healthy controls (Other): healthy controls
  Interventions: Diagnostic Test: histologic evaluation; Diagnostic Test: biochemical analysis; Diagnostic Test: clinical examination
- patients having OPMDs with dysplasia (Other): patients having OPMDs with dysplasia
  Interventions: Diagnostic Test: histologic evaluation; Diagnostic Test: biochemical analysis; Diagnostic Test: clinical examination
- patients having OPMDs without dysplasia (Other): patients having OPMDs without dysplasia
  Interventions: Diagnostic Test: histologic evaluation; Diagnostic Test: biochemical analysis; Diagnostic Test: clinical examination
- oral cancer patients (Other): oral cancer patients
  Interventions: Diagnostic Test: histologic evaluation; Diagnostic Test: biochemical analysis; Diagnostic Test: clinical examination

INTERVENTIONS:
Diagnostic Test: histologic evaluation — histologic evaluation
Diagnostic Test: biochemical analysis — IL-6, IL-8 and sCD44
Diagnostic Test: clinical examination — clinical examination

SUMMARY:
The present investigation was conducted on 100 individuals allocated into four groups; 25 healthy controls, 25 patients having OPMDs with dysplasia; 25 patients having OPMDs without dysplasia, and 25 oral cancer patients. Demographic data including data related to different risk factors, modified gingival index, oral hygiene level, in addition to salivary levels of IL-6, IL-8 and sCD44 were assessed.

DETAILED DESCRIPTION:
Histopathologic evaluation:

Biopsy samples were obtained from all lesions to verify the diagnosis and establish the presence of dysplasia in the potentially premalignant lesions before allocating patients to their specific groups.

History and clinical assessment:

Demographic data as age and gender, medical history and habits as smoking and alcohol were obtained during patient interview. Modified gingival index (MGI), level of oral hygiene (OH) and the number of remaining natural teeth were also assessed. Subjects not willing to sign a written informed consent, pregnant females, lactating mothers, and patients with immunosuppressive disorders were excluded.

Modified gingival index (MGI) evaluates the presence and degree of gingival inflammation. A score of 0 means absence of inflammation. 1 indicates mild inflammation (slight redness) of any part of the gingiva. 2- mild inflammation of the whole gingiva. 3- moderate inflammation (moderate redness, edema, and/or hypertrophy) of the gingiva. 4-severe inflammation (marked redness and spontaneous bleeding) of the gingiva. Level of OH care was evaluated corresponding to the OH habits of the patient and efficiency of plaque removal. OH, level is scored as: 1- very good, 2- good, 3- fair, and 4- poor OH.

Collection of 1.0-2.0 mL of whole unstimulated saliva was obtained between nine and twelve in the morning, to evade diurnal alteration. Participants refrained from eating, smoking, brushing, and mouthwash use, 2 hours before to salivary sampling, which were stored at -70 ◦C till analyzed.

Quantification of salivary IL-6, IL-8, and sCD44 in all samples using an ELISA kit

List of abbreviations:

OSCC: Oral squamous cell carcinoma OPMDs: Oral potentially malignant disorders HNSCC: Head and neck squamous cell carcinoma MGI: Modified gingival index. OH: Level of oral hygiene ROC: Receiver operating characteristic

ELIGIBILITY:
Inclusion Criteria:

* patients above 18 years both males and females patients presenting with OPMDs

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2023-07-15 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-15 (Actual)

PRIMARY OUTCOMES:
Quantities of IL-6 and IL-8 | baseline
  assessed in all samples using an ELISA kit (Orgenium laboratories, Business Unit, Finland). The test principles apply a sandwich-type ELISA where a polyclonal anti-antibody, adsorbed onto microwells, binds IL-6 and IL-8 in the samples, Results were expressed in pg/ml
Levels of sCD44 | Baselone
  measured using an ELISA assay (Bender MedSystems, Vienna, Austria) that identifies all normal and variant isoforms. Saliva samples were centrifuged at 2000 Xg and the supernatants were separated and stored at -80 ̊C till processing, which was done according to manufacturer's instructions. Results were expressed in ng/ml.

SECONDARY OUTCOMES:
MGI (modified gingival index) | baseline
  Modified gingival index (MGI) evaluates the presence and degree of gingival inflammation. A score of 0 means absence of inflammation. 1 indicates mild inflammation (slight redness) of any part of the gingiva. 2- mild inflammation of the whole gingiva. 3- moderate inflammation (moderate redness, edema, and/or hypertrophy) of the gingiva. 4-severe inflammation (marked redness and spontaneous bleeding) of the gingiva.

CONTACTS AND LOCATIONS:
Locations (1):
- British University in Egypt, Cairo, Egypt